CLINICAL TRIAL: NCT03422081
Title: Validation of the Dosage of Asymmetric Dimethylarginine (ADMA) Plasma in the Assessment of Endothelial Dysfunction During Growth Hormone Deficiency and Intrauterine Growth Retardation
Brief Title: Growth and Asymmetric diMethylArginine
Acronym: GAMMA
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2012_61; 2013-A00830-45 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-01-10; First posted 2018-02-05 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Growth Hormone Deficiency; Small-for-gestational Age
Keywords: endothelial dysfunction; doppler ultrasound examination; nitric oxide
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- growth hormone deficiency
  Interventions: Diagnostic Test: arterial doppler ultrasound
- small for gestational age
  Interventions: Diagnostic Test: arterial doppler ultrasound
- matched controls
  Interventions: Diagnostic Test: arterial doppler ultrasound

INTERVENTIONS:
Diagnostic Test: arterial doppler ultrasound — doppler ultrasound

SUMMARY:
Principal objective : Validation of a handy biochemical parameter, plasma concentration of Asymmetric DimethylArginine (ADMA), based on a recognize biochemical parameter, the dilation of the brachial artery, at ultrasound examination, after the deflation of a cushion to evaluate artery dysfunction (vascular suffering) in growth diseases, growth hormone deficiency (GHD) and intrauterine growth retardation (IUGR)

Secondary objectives:

* Comparison of ADMA plasma concentrations with dose of matched healthy control children
* Investigation of the mechanisms of arterial dysfunction, inflammation, oxidative stress and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Group A: GHD, defined by 2 GH peaks less than 6.6 ng/ml (20 mU/L) at two stimulation tests
* Group B: IUGR, defined by a birth length and/or a birth weight inferior to - 2 SD for gestational age according to Usher and McLean charts
* Group C: Control children matched to children matched to subjects of groups A and B, according to gender and age
* Informed consent signed by representative of the parental authority

Exclusion Criteria:

* Chronic disabling disease (ex: diabetes, severe asthma)
* Evolving cancer
* Severe psychiatric disorder (ex: autism, schizophrenia; severe depression)
* Hypothalamic tumor (ex: craniopharyngioma)
* Anamnesis of cranial irradiation
* Overweight, obesity or thinness
* Precocious puberty
* Non-replacing therapy by glucocorticoids or sex steroids less than 1 month before the exploration
* Anterior treatment by recombinant human GH
* Other conditions, treatments or habits impacting arterial reactivity: acrocyanosis, cryoglobulinemia, beta adrenergic blocking habits, tobacco smoking or other drug addictions, dyslipidemia
* Pregnancy or lactation
* Acute infection less than three weeks before the investigation
* Participation to a therapeutic protocol
* Impossibility for the representatives of the parental authority to understand the objectives of the protocol
* Absence of social security coverage. Refusal by the parents to sign the informed consent or oral refusal by the child to participate to the study

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric patients with growth disorders and matched control children
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Plasma Asymmetric Dimethylarginine (ADMA) | At baseline
  Correlation between ADMA (Asymmetric DimethylArginine, a collateral derivate of nitric oxide metabolism) levels and the percentage of dilation of the brachial artery at Doppler ultrasound examination.
  The dosage will be performed by high pressure liquid chromatography followed by tandem mass spectrometry (HPLC-MS / MS)
Percentage of dilation of the brachial artery at Doppler ultrasound examination. | At baseline.
  Correlation between ADMA (Asymmetric DimethylArginine, a collateral derivate of nitric oxide metabolism) levels and the percentage of dilation of the brachial artery at Doppler ultrasound examination.

SECONDARY OUTCOMES:
Difference of ADMA concentration between the patient and the control groups | At baseline
Correlation of ADMA levels with diverse cardiovascular risk factors | At baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Weill, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (2):
- France (2):
  - Hôpital Jeanne de Flandre - CHRU de Lille, Lille
  - CHU Purpan, Toulouse

IPD SHARING:
Plan to Share IPD: No